CLINICAL TRIAL: NCT00680615
Title: QuitSpit: An Internet-Based Smokeless Tobacco Cessation Program for Teens
Brief Title: An Internet-Based Smokeless Tobacco Cessation Program for Teens
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01CA118575 (NIH)
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Smokeless Tobacco Use
Keywords: Smokeless tobacco
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (Experimental)
  Interventions: Behavioral: Usual Care
- Enhanced (Experimental)
  Interventions: Behavioral: Tailored, enhanced condition

INTERVENTIONS:
Behavioral: Tailored, enhanced condition — Intervention will provide a personalized, interactive tobacco cessation Web application, based on existing empirically validated smokeless tobacco cessation programs.
  Arms: Enhanced
Behavioral: Usual Care — The Usual Care condition will provide access to typical smokeless tobacco cessation information and links to commonly available Web-based smokeless tobacco cessation resources.
  Arms: Usual Care

SUMMARY:
To compare the efficacy of a targeted, tailored, and highly interactive smokeless tobacco cessation website to a website with more static information that is similar to websites that can be found through a typical Internet search.

ELIGIBILITY:
Inclusion Criteria:

* 14-25 years of age
* Have access to the Internet
* Currently using smokeless tobacco products
* Currently contemplating quitting all tobacco products
* Able to read and write English; and
* Willing to share phone number, e-mail, and mailing address with the research project

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1716 (Actual)
Dates: Start 2008-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Abstinence from all tobacco | 3 months and 6 months
Abstinence from smokeless tobacco | 3 months and 6 months

SECONDARY OUTCOMES:
Evaluate the relative effectiveness of the two programs on secondary outcomes, including reduction in smokeless tobacco use, number of quit attempts, and confidence in quitting. | 3 months and 6 months
Identify participant characteristics, including demographic characteristics, initial smokeless tobacco use and dependence, and patterns of program use that predict treatment outcomes. | 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Herbert H. Severson, PhD, Principal Investigator — Oregon Research Institute; Brian G Danaher, PhD, Principal Investigator — Oregon Research Institute
Locations (1):
- Oregon Research Institute, Eugene, Oregon, United States